CLINICAL TRIAL: NCT06406985
Title: Developing a Weight Management Class as Curriculum for Rural Illinois Extension Nutrition Educators and as a Reach-Out Tool for an Online Weight Loss Program to Rural Residents
Brief Title: Developing a Weight Management Class as a Recruitment Tool for an Online Weight Loss Program to Rural Illinois Residents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB24-0474
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EMPOWER Weight-Loss Participants (Experimental): All weight-loss participants will receive the same protocol and weight-loss education materials. Nutrition coaching is individualized to participant needs, but emphasizes the program's core themes throughout.
  Interventions: Behavioral: Weight-loss through dietary and lifestyle changes

INTERVENTIONS:
Behavioral: Weight-loss through dietary and lifestyle changes — Weight-loss participants will complete one online, self-paced education session each week for 12 weeks. Education sessions focus on topics such as self-monitoring weight, meal routines, and dietary habits with an emphasis on protein and fiber intake. During these 12 weeks, participants will receive weekly messages from nutrition coaches as well as a monthly nutrition coaching call. After the first 12 weeks, participants will enter a follow-up period where nutrition coaching messaging will occur as needed and with the opportunity to still participate in a monthly nutrition coaching call. Participants are asked to weigh daily on a provided WiFi scale that automatically uploads their weight data to a website for researchers and coaches to monitor. Participants will also submit food records and self-reported weight and hip circumferences.

SUMMARY:
The purpose of this study is to identify how to maintain a sustainable collaboration Illinois Extension Nutrition and Wellness Educators while continuing to offer an online weight-loss program, EMPOWER, to rural Illinois residents.

* The primary aim of the study is to determine if an Extension-delivered introductory weight management class will be successful in recruiting rural individuals interested in losing weight to the EMPOWER weight-loss program.
* The secondary aim is to enroll interested rural participants in an online weight loss intervention that focuses on promoting dietary and lifestyle behavioral changes to achieve ≥5 percent weight loss.

Participants who participate in the EMPOWER weight-loss intervention will:

1. Complete 12 online educational sessions over a 3-month period followed by a 9-month follow-up period.
2. Participate in daily self-weighing using a provided WiFi-enabled scale.
3. Will have a monthly nutrition coaching call once per month for the 12-month duration of the study.
4. Will complete food records and self-report waist and hip circumference measures at baseline, 3-months, and 12-months.

DETAILED DESCRIPTION:
The purpose of the investigators' study is to identify how to maintain a sustainable collaboration with the investigator-developed weight-loss program, EMPOWER, and rural Illinois Extension Nutrition and Wellness Educators. The investigators are aiming to identify potential barriers of recruitment, rolling enrollment, and intervention methods to enhance the success of maintaining this collaboration at a distance and continue to offer weight management services to rural areas. If the investigators can demonstrate continual, successful collaboration with the Extension educators, they can work towards expanding EMPOWER to even more communities. In objective 1, the investigators will create an introductory weight management curriculum in collaboration with three Illinois Extension nutrition and wellness educators that can be disseminated to their respective rural populations (Christian, Jersey, Macoupin, Montgomery, Jo-Daviess, Stephenson, Clark, Crawford, and Edgar counties). The class will also be supplemented with healthy recipe handouts. The class serves to fulfill curricula requirements for Extension educators in the area of chronic disease prevention and management while simultaneously serving as a recruitment method for the investigators' EMPOWER program. This objective serves to answer the research question of whether offering a weight management class through Extension is a feasible way to recruit those in need of weight-loss to EMPOWER while maintaining long-term collaboration with Extension. The data obtained from this objective includes an exit interview with each of the Extension educators, the number of attendees from each Extension class, as well as an optional survey provided to the Extension class attendees. No identifiable information will be obtained from the Extension class attendees unless they express interest in the study recruitment flyer and proceed to fill out an eligibility form. Objective 2 of the study is to enroll interested rural participants into a 3-month intervention and 9- month follow-up EMPOWER weight loss trial with statistically significant weight loss being the expected outcome at the end of the 12 months. EMPOWER is an online weight-loss program that aims to achieve safe weight-loss through sustainable dietary and lifestyle changes. Participants of EMPOWER will be provided online educational materials through Illinois eText and nutrition coaching from registered dietitians and nutrition students via email/messaging correspondence and monthly phone/video calls. Participants will be asked to self-weigh everyday as a method to monitor energy balance. MealPlot, a web- application developed by the investigators, will be available for participants to submit food records, message their coach, see their weight data, and monitor their protein and fiber intake. Overall, successful EMPOWER recruitment from the Extension class and following success of EMPOWER enrollees losing statistically significant weight would lead to an improvement of health among rural residents where weight care strategies are typically limited and would demonstrate the feasibility of long-term collaboration with Extension educators.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than or equal to 28 kg/m^2
* age 18-75
* ability to access the internet and smartphone
* fluent in English
* having primary residence in a rural Illinois county

Exclusion Criteria:

* Pregnant or lactating
* previous or planned bariatric surgery
* BMI less than 28 kg/m^2
* Age less than 18 or greater than 75
* no access to internet and smartphone/smart device
* on GLP-1 Receptor Agonist weight loss medication
* Diagnosed with an eating disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment feasibility | 3 months
  Recruitment Goal: Recruitment will be completed within 3-months and 50% or more of submitted eligibility forms will be from those who attended the introductory weight-management class with Extension.
Sustainability of collaboration | end of 12-month study
  Exit interviews will be conducted with collaborators to identify themes surrounding the nature of the collaboration.

SECONDARY OUTCOMES:
Weight-loss | end of 12-month study
  Weight-loss of greater than or equal to 5 percent total body weight when compared to baseline in each participant.
Dietary change | end of 12-month study
  Statistically significant increase in dietary protein and fiber density (grams/100 kilocalories) when compared to baseline 3-day food records.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: EMPOWER Study Website — https://publish.illinois.edu/empower-uiuc/